CLINICAL TRIAL: NCT00403767
Title: A Prospective, Randomized, Double-Blind, Parallel-Group, Multicenter, Non-inferiority Study Comparing the Efficacy and Safety of Rivaroxaban (BAY 59-7939) With Warfarin for the Prevention of Stroke and Non-Central Nervous System Systemic Embolism in Subjects With Non-Valvular Atrial Fibrillation
Brief Title: An Efficacy and Safety Study of Rivaroxaban With Warfarin for the Prevention of Stroke and Non-Central Nervous System Systemic Embolism in Patients With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR012157; 39039039AFL3001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); ROCKET AF (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2006-004595-13 (EudraCT Number)
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation; Stroke; Embolism
Keywords: Atrial Fibrillation; Stroke; Embolism; Non-central nervous system systemic embolism; Non-valvular atrial fibrillation; Blood Clot; Rivaroxaban; Warfarin; Anticoagulants; Arrhythmias, Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Embolism; Thrombosis; Arrhythmias, Cardiac | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban; Drug: Matching placebo for Rivaroxaban arm (Warfarin placebo)
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin; Drug: Matching placebo for Warfarin arm (Rivaroxaban placebo)

INTERVENTIONS:
Drug: Rivaroxaban — Type=exact number, unit=mg, number=20, form=tablet, route=oral use. One 20 mg tablet once daily for an expected maximum treatment period of up to 32 months that may extend up to 4 years (Patients with moderate renal impairment at screening willl have a dose adaptation to rivaroxaban 15 mg, orally, once daily for an expected maximum treatment period of up to 32 months that may extend up to 4 years)
  Arms: Rivaroxaban
Drug: Warfarin — Type=exact number, unit=mg, number=1, 2.5, or 5 mg, form=tablet, route=oral use. Number of warfarin tablets to be determined based on target INR values once daily for an expected maximum treatment period of up to 32 months that may extend up to 4 years
  Arms: Warfarin
Drug: Matching placebo for Rivaroxaban arm (Warfarin placebo) — Form=tablet, route=oral. One warfarin placebo tablet taken orally once daily for up to an expected maximum treatment period of 32 months that may extend up to 4 years
  Arms: Rivaroxaban
Drug: Matching placebo for Warfarin arm (Rivaroxaban placebo) — Form-tablet, Route=oral administration. Number of rivaroxaban placebo determined by the number of warfarin tablets taken. Duration of treatment is up to an expected maximum treatment period of 32 months that may extend up to 4 years
  Arms: Warfarin

SUMMARY:
The purpose of this study is to compare the efficacy and safety of rivaroxaban with warfarin for the prevention of blood clots in the brain (referred to as stroke) and blood clots in other parts of the body referred to as non-central nervous system systemic embolism) in patients with non-valvular atrial fibrillation (a heart rhythm disorder).

DETAILED DESCRIPTION:
Patients with non-valvular atrial fibrillation who are at risk for stroke and non-central nervous system (non-CNS) systemic embolism, will be randomized (assigned by chance) to receive treatment with rivaroxaban or warfarin, two different anticoagulants (substances that prevent blood clots). Treatment will be double-blinded (neither the patient nor study staff will know which study drug is assigned to patients during the study). Patients assigned to rivaroxaban will receive rivaroxaban 20 mg orally (p.o.) once daily (OD) plus warfarin placebo p.o. OD titrated to a target sham international normalized ratio (INR) of 2.5. Patients with moderate renal impairment at screening will receive rivaroxaban 15 mg p.o. OD. Patients assigned to warfarin will receive warfarin p.o. OD titrated to a target INR of 2.5 plus rivaroxaban placebo p.o. OD. The maximum expected length of treatment is up to 32 months but may be extended up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented atrial fibrillation on 2 separate occasions within 6 months before screening
* History of a prior stroke, transient ischemic attack or non-neurologic systemic embolism believed to be cardiac in origin, or at least two of the following risk factors: heart failure, hypertension, age 75 years or greater, diabetes mellitus

Exclusion Criteria:

* Significant mitral stenosis
* Transient atrial fibrillation caused by a reversible disorder
* Active internal bleeding
* Severe disabling stroke
* History of intracranial bleeding
* Hemorrhagic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14269 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (932):
- United States (295):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Geneva, Alabama
  - Mobile, Alabama
  - Pell City, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Fort Smith, Arkansas
  - Little Rock, Arkansas
  - Anaheim, California
  - Bakersfield, California
  - Carmichael, California
  - Corona, California
  - Fair Oaks, California
  - Glendale, California
  - Healdsburg, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Mission Viejo, California
  - Modesto, California
  - Mountain View, California
  - Northridge, California
  - Oakland, California
  - Orange, California
  - Pismo Beach, California
  - Sacramento, California
  - San Diego, California
  - San Leandro, California
  - Santa Clara, California
  - Santa Monica, California
  - Santa Rosa, California
  - Sylmar, California
  - Torrance, California
  - Ventura, California
  - Yuba City, California
  - Boulder, Colorado
  - Denver, Colorado
  - Littleton, Colorado
  - Pueblo, Colorado
  - Danbury, Connecticut
  - Guilford, Connecticut
  - Newark, Delaware
  - Bradenton, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - DeBary, Florida
  - Deerfield Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Fort Walton Beach, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Hudson, Florida
  - Inverness, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Largo, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Ocala, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Palm Beach Gardens, Florida
  - Palm Harbor, Florida
  - Port Charlotte, Florida
  - Safety Harbor, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Nampa, Idaho
  - Aurora, Illinois
  - Bannockburn, Illinois
  - Chicago, Illinois
  - Evergreen Park, Illinois
  - Fulton, Illinois
  - Lombard, Illinois
  - Melrose Park, Illinois
  - Moline, Illinois
  - Park Ridge, Illinois
  - Peoria, Illinois
  - Quincy, Illinois
  - Rock Island, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Watseka, Illinois
  - Anderson, Indiana
  - Hammond, Indiana
  - Indianapolis, Indiana
  - Merrillville, Indiana
  - Muncie, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Waterloo, Iowa
  - Crestview Hills, Kentucky
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Mount Sterling, Kentucky
  - Owensboro, Kentucky
  - Houma, Louisiana
  - Lake Charles, Louisiana
  - New Orleans, Louisiana
  - Thibodaux, Louisiana
  - Vidalia, Louisiana
  - Bangor, Maine
  - Scarborough, Maine
  - Annapolis, Maryland
  - Beltsville, Maryland
  - Columbia, Maryland
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Brighton, Massachusetts
  - Framingham, Massachusetts
  - Bay City, Michigan
  - Bridgman, Michigan
  - Chelsea, Michigan
  - Dearborn, Michigan
  - Detroit, Michigan
  - Lansing, Michigan
  - Mount Clemens, Michigan
  - Petoskey, Michigan
  - Traverse City, Michigan
  - Troy, Michigan
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Picayune, Mississippi
  - Tupelo, Mississippi
  - Lexington, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Anaconda, Montana
  - Great Falls, Montana
  - Beatrice, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Pahrump, Nevada
  - Manchester, New Hampshire
  - Bridgewater, New Jersey
  - Elmer, New Jersey
  - Haddon Heights, New Jersey
  - New Brunswick, New Jersey
  - Paterson, New Jersey
  - Ridgewood, New Jersey
  - Sewell, New Jersey
  - Springfield, New Jersey
  - Toms River, New Jersey
  - Wayne, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Buffalo, New York
  - Cortlandt Manor, New York
  - East Syracuse, New York
  - New York, New York
  - Northport, New York
  - Saratoga Springs, New York
  - Schenectady, New York
  - Staten Island, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Williamsville, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Hickory, North Carolina
  - Jacksonville, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Reidsville, North Carolina
  - Rocky Mount, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Minot, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Fairfield, Ohio
  - Mansfield, Ohio
  - Massillon, Ohio
  - Maumee, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Bartlesville, Oklahoma
  - Midwest City, Oklahoma
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Doylestown, Pennsylvania
  - Jeannette, Pennsylvania
  - Jersey Shore, Pennsylvania
  - Lansdale, Pennsylvania
  - Leetsdale, Pennsylvania
  - Lewistown, Pennsylvania
  - Norristown, Pennsylvania
  - North Wales, Pennsylvania
  - Philadelphia, Pennsylvania
  - Philipsburg, Pennsylvania
  - Phoenixville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sayre, Pennsylvania
  - Scranton, Pennsylvania
  - Shippensburg, Pennsylvania
  - State College, Pennsylvania
  - Topton, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Wormleysburg, Pennsylvania
  - Wyomissing, Pennsylvania
  - Pawtucket, Rhode Island
  - Westerly, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Easley, South Carolina
  - Sumter, South Carolina
  - Rapid City, South Dakota
  - Athens, Tennessee
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Harriman, Tennessee
  - Jackson, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Lexington, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Beaumont, Texas
  - Brownsville, Texas
  - Corpus Christi, Texas
  - Daingerfield, Texas
  - Dallas, Texas
  - DeSoto, Texas
  - Fort Sam Houston, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Humble, Texas
  - Hurst, Texas
  - Kerrville, Texas
  - Kingwood, Texas
  - Lubbock, Texas
  - McAllen, Texas
  - Odessa, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tomball, Texas
  - Victoria, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Blacksburg, Virginia
  - Chester, Virginia
  - Danville, Virginia
  - Fairfax, Virginia
  - Fredericksburg, Virginia
  - Lynchburg, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Williamsburg, Virginia
  - Bellingham, Washington
  - Port Orchard, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - Burlington, Wisconsin
  - Elkhorn, Wisconsin
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
  - Wausau, Wisconsin
- Argentina (13):
  - Bahía Blanca
  - Buenos Aires
  - Cipolletti
  - Corrientes
  - Córdoba
  - La Plata
  - Mar del Plata
  - Quilmes
  - Rosario
  - Salta
  - San Martín
  - San Miguel de Tucumán
  - Santa Fe
- Australia (30):
  - Adelaide
  - Auchenflower
  - Bedford Park
  - Box Hill
  - Caboolture
  - Cairns
  - Camperdown
  - Chermside
  - Clayton
  - Coffs Harbour
  - Footscray
  - Garran
  - Geelong
  - Gosford
  - Heidelberg Heights
  - Herston
  - Hobart
  - Joondalup
  - Lismore
  - Liverpool
  - Miranda
  - Nedlands
  - New Lambton Heights
  - Parkville
  - Penrith
  - Prahran
  - Reservoir
  - Southport
  - Windsor
  - Wolloongabba
- Austria (5):
  - Feldkirch Vorarlberg Vorarlber
  - Graz
  - Tulln Niederosterreich Niedero
  - Vienna
  - Wien Wien
- Belgium (14):
  - Antwerp
  - Bonheiden
  - Brasschaat
  - Bruges
  - Brussels
  - Ghent
  - Haine-Saint-Paul
  - Leuven
  - Mol
  - Nivelles
  - Ottignies
  - Roeselare
  - Seraing
  - Tienen
- Brazil (23):
  - Belo Horizonte
  - Blumenau
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Campo Grande
  - Curitiba
  - Fortaleza
  - Goiânia
  - Maceió
  - Maringá
  - Marília
  - Porto Alegre
  - Recife
  - Rio de Janeiro
  - Rio de Janeiro Br
  - Salvador
  - Santo André
  - São Caetano do Sul
  - São José do Rio Preto
  - São Paulo
  - Sorocaba
  - Uberlândia
- Bulgaria (6):
  - Dimitrovgrad
  - Pleven
  - Plovdiv
  - Russel
  - Sofia
  - Veliko Tarnovo
- Canada (70):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbotsford, British Columbia
  - Burnaby, British Columbia
  - Campbell River, British Columbia
  - Delta, British Columbia
  - Kelowna, British Columbia
  - Langley, British Columbia
  - New Westminster, British Columbia
  - Penticton, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - West Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Sydney, Nova Scotia
  - Ajax, Ontario
  - Beamsville, Ontario
  - Belleville, Ontario
  - Brampton, Ontario
  - Burlington, Ontario
  - Cambridge, Ontario
  - Corunna, Ontario
  - Courtice, Ontario
  - E. London, Ontario
  - Etobicoke, Ontario
  - Fort Erie, Ontario
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Listowel, Ontario
  - London, Ontario
  - Markham, Ontario
  - Mississauga, Ontario
  - North Bay, Ontario
  - North York, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Parry Sound, Ontario
  - Richmond Hill, Ontario
  - Sarnia, Ontario
  - Sault Ste. Marie, Ontario
  - Scarborough Village, Ontario
  - Strathroy, Ontario
  - Thornhill, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Whitby, Ontario
  - York, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Joliette, Quebec
  - Jonquière, Quebec
  - Lachine, Quebec
  - Longueuil, Quebec
  - Mirabel, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Saint-Jérôme, Quebec
  - Saint-Lambert, Quebec
  - Saint-Léonard, Quebec
  - Sherbrooke, Quebec
  - North Battleford, Saskatchewan
  - Saskatoon, Saskatchewan
- Chile (12):
  - Arica I Region
  - Chila
  - Concepción VIII
  - Osorno X Region
  - Osorno X Región
  - Rancagua VI Region
  - San Felipe V Region
  - Santiago de Chile Rm
  - Santiago Rm
  - Temuco IX
  - Valdivia X Región
  - Viña Del Mar V Región
- China (20):
  - Beijing
  - Changchun
  - Changsha
  - Changzhou
  - Chengdu
  - Chongqing
  - Dalian
  - Daqing
  - Guangzhou
  - Haikou
  - Hangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Shanghai
  - Shenyang
  - Suzhou
  - Tianjin
  - Wuhan
  - Xi'an
- Colombia (11):
  - Barranquilla
  - Barranquilla Atlántico Atlanti
  - Bogota D C
  - Bogota Dc
  - Bogotá Dc Dc
  - Bogotá Dc
  - Cali Valle Del Cauca
  - Cali Valley Del Cauca
  - Medellin Antioquia
  - Medellín
  - Santander
- Czechia (18):
  - Brno
  - Chomutov
  - Hradec Králové
  - Kutná Hora
  - Liberec
  - Litomyšl
  - Náchod
  - Olomouc
  - Ostrava
  - Pardubice
  - Prague
  - Praha 10 N/A
  - Ráj
  - Slaný
  - Svitavy
  - Trutnov
  - Uherské Hradistì 6
  - Zlín
- Denmark (12):
  - Copenhagen
  - Elsinore
  - Esbjerg
  - Frederiksberg
  - Gentofte Municipality
  - Hellerup
  - Hvidovre
  - Koege
  - Næstved
  - Roskilde
  - Slagelse
  - Viborg
- Finland (6):
  - Helsinki
  - Jyväskylä
  - Kuopio
  - Mikkeli
  - Oulu
  - Turku
- France (24):
  - Albi
  - Arras
  - Bayonne
  - Belfort
  - Besançon
  - Béziers Languedoc-Roussillon
  - Bourg-en-Bresse
  - Brest
  - Carcassonne
  - Clermont-Ferrand
  - Corbeil-Essonnes
  - Lille
  - Marseille
  - Montbéliard
  - Montpellier
  - Paris
  - Perpignan
  - Poitiers
  - Saint-Brieuc
  - Saint-Jean-de-Verges
  - Strasbourg
  - Thionville
  - Toulouse
  - Trélivan
- Germany (62):
  - Aalen
  - Berlin
  - Berlin/Spandau
  - Biberach
  - Bochum
  - Bonn
  - Chemnitz
  - Coburg
  - Dachau
  - Dortmund
  - Dresden
  - Duisburg
  - Ebersbach
  - Eilenburg
  - Erfurt
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Greifswald
  - Halle
  - Hamburg
  - Hartmannsdorf
  - Heidelberg
  - Henstedt-Rhen
  - Herford
  - Homburg/Saar
  - Jena
  - Jülich
  - Kamen
  - Karlsbad
  - Kassel
  - Kirchzarten
  - Krefeld
  - Leipzig
  - Ludwigsburg
  - Ludwigshafen
  - Lüneburg
  - Magdeburg
  - Mainz
  - Mannheim
  - Markkleeberg
  - Meißen
  - Melsungen
  - Mönchengladbach
  - Mühldorf
  - Mülheim
  - München
  - Münster
  - Neuwied
  - Nienburg
  - Nuremberg
  - Paderborn
  - Potsdam
  - Riesa
  - Rottweil
  - Sachsen
  - Siegen
  - Ulm
  - Wermsdorf
  - Witten
  - Wolmirstedt
  - Wuppertal
- Greece (7):
  - Athens Attica
  - Ioannina
  - Maroussi Athens
  - Pátrai
  - Piraeus Attica
  - Tripoli
  - Voula Attica
- Hong Kong (4):
  - Aberdeen
  - Hong Kong
  - Kln
  - Shatin
- Hungary (15):
  - Budapest
  - Budapest Nap
  - Debrecen County
  - Eger
  - Gyõr
  - Gyöngyös
  - Kesckemet
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Szombathely
  - Veszprém
  - Zalaegerszeg
- India (18):
  - Ahmedabad
  - Bangalore
  - Bikaner
  - Chennai
  - Coimbatore
  - Gandhinagar Guiarat
  - Hyderabad
  - Hyderabad Andra Pradesh
  - Jalandhar
  - Madurai
  - Mangalore
  - Mumbai
  - Mysore
  - New Delhi
  - Pune
  - Sūraj
  - Vadodara
  - Visakhapatnam
- Israel (15):
  - Afula
  - Ashkelon
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Nazareth
  - Netanya
  - Petah Tikva
  - Poria – Neve Oved
  - Rehovot
  - Safed
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Malaysia (3):
  - Kelantan
  - Kuala Lumpur
  - Sarawak
- Mexico (11):
  - Aguascalientes
  - Culiacán Sinaloa/Mèxico
  - Guadalajara
  - Hermosillo
  - Mexico City
  - Monterrey
  - Monterrey Nuevo Leòn
  - Querétaro
  - San Luis Potosí City
  - Sinaloa
  - Zapopan
- Netherlands (21):
  - 's-Hertogenbosch
  - Alkmaar
  - Amersfoort
  - Amsterdam
  - Blaricum
  - Delft
  - Gc Tilburg
  - Gouda
  - Groningen
  - Haarlem
  - Heerlen
  - Hoofddorp
  - Hoorn
  - Leeuwarden
  - Leidschendam
  - Maastricht
  - Meppel
  - Nijmegen
  - Schiedam
  - The Hague
  - Veldhoven
- New Zealand (6):
  - Christchurch
  - Dunedin
  - Grafton
  - Hamilton
  - Takapuna Auckland
  - Wellington
- Norway (12):
  - Ålesund
  - Bergen
  - Elverum
  - Hamar
  - Jessheim
  - Lillehammer
  - Moss
  - Oslo
  - Sandefjord
  - Sandnes
  - Sandvika
  - Skedsmokorset
- Peru (3):
  - L41 Lima Lima
  - Lima
  - Lima 1 Lima Lima
- Philippines (5):
  - Cebuu City
  - Davao City
  - Iloilo City
  - Manila
  - Quezon City
- Poland (25):
  - Bydgoszcz
  - Gdansk
  - Gdynia
  - Katowice
  - Katowice-Ochojec
  - Krakow
  - Lodz
  - Olsztyn
  - Opole
  - Ostrowiec
  - Oława
  - Piotrkow Trybunalski
  - Poznan
  - Płock
  - Siedlce
  - Sieradz
  - Skierniewice
  - Starogard Gdanski Nap
  - Szczecin
  - Szczecin Nap
  - Torun
  - Warsaw
  - Wroclaw
  - Włocławek
  - Żyrardów
- Romania (10):
  - Brasov
  - Bucharest
  - Craiova
  - Focşani
  - Iași
  - Oradea
  - Sibiu
  - Suceava
  - Tg Mures
  - Timișoara
- Russia (20):
  - Barnaul
  - Chelyabinsk
  - Chelyabinsk Chelyabinsk Region
  - Kemerovo
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Novosibirsk Nap
  - Orenburg
  - Perm
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tomsk
  - Tyumen Tyumen Region
  - Yaroslavl
  - Yaroslavl Nap
  - Yekaterinburg
- Singapore, Singapore
- South Africa (13):
  - Bloemfontein Free State
  - Bloemfontein Orange Free State
  - Cape Town
  - Cape Town Western Cape
  - Centurion Gauteng
  - Durban Kwa Zulu Natal
  - Johannesburg Gauteng
  - Kempton Park Gauteng
  - Port Elizabeth Eastern Cape
  - Pretoria Gauteng
  - Somerset West Western Cape
  - Vanderbijlpark
  - Worcester Western Cape
- South Korea (9):
  - Anyang
  - Daegu
  - Daejeon
  - Goyang
  - Kyonggi-Do
  - Pusan
  - Seoul
  - Sungnam
  - Suwon
- Spain (20):
  - A Coruña
  - Alicante
  - Almería
  - Baracaldo Vizcaya
  - Barcelona
  - Burgos
  - Guadalajara
  - La Corona
  - Madrid
  - Málaga
  - Oviedo
  - Palma de Mallorca
  - Pamplona
  - Pontevedra
  - Sabadell
  - San Sebastián Guipúzcoa
  - Seville
  - Terrassa
  - Valencia
  - Valladolid
- Sweden (5):
  - Ljungby
  - Lund
  - Sala
  - Skövde
  - Uppsala
- Switzerland (4):
  - Basel Bs
  - Bruderholz
  - Geneva
  - Zurich
- Taiwan (7):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Tamshui
  - Taoyuan District
- Thailand (6):
  - Bangkok
  - Bangkok Noi
  - Chiang Mai
  - Pathum Thani
  - Phathumwan
  - Ratchatewi
- Turkey (Türkiye) (16):
  - Adana
  - Ankara
  - Antalya
  - Aydin
  - Denizli
  - Diyarbakır
  - Eskişehir
  - Görükle
  - Istanbul
  - Izmir
  - İzmit
  - Kayseri
  - Konya
  - Malatya Nap
  - Mersin
  - Samsun
- Ukraine (22):
  - Cherkassy
  - Chernihiv
  - Dnipro
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kirovograd
  - Kyiv
  - Luhansk
  - Lviv
  - O1103 Kyiv
  - Odesa
  - Poltava
  - Simferopil
  - Sumy
  - Ternopil
  - Uzhhorod
  - Vinnitsya
  - Vinnytsia
  - Zaporizhzhya
  - Zhytomyr
- United Kingdom (25):
  - Aberdeen
  - Belfast
  - Birmingham
  - Bournemouth
  - Cambridgeshire
  - Chelmsford
  - Chesterfield
  - Colchester
  - Craigavon
  - Devon
  - Dundee
  - Glasgow
  - Harrogate
  - Hull
  - Leicester
  - Lincoln
  - Liverpool
  - London
  - Nottingham
  - Plymouth
  - Romford
  - Sheffield
  - Stirling
  - Stoke-on-Trent
  - York
- Venezuela (3):
  - Caracas
  - Maracaibo Estado Zulia
  - Maracay Estado Aragua

REFERENCES:
- [Derived] Dobesh PP, Volkl AA, Pap AF, Damaraju CV, Levitan B, Yuan Z, Amin AN. Benefit-Risk Assessment of Rivaroxaban in Older Patients With Nonvalvular Atrial Fibrillation or Venous Thromboembolism. Drugs Aging. 2025 May;42(5):469-484. doi: 10.1007/s40266-025-01192-7. Epub 2025 Mar 31. PMID 40163217
- [Derived] Ungar L, Rodriguez F, Hellkamp AS, Becker RC, Berkowitz SD, Breithardt G, Fox KAA, Hacke W, Halperin JL, Hankey GJ, Nessel CC, Singer DE, Patel MR, Piccini JP, Mahaffey KW. Patient-Reported Satisfaction and Study Drug Discontinuation: Post-Hoc Analysis of Findings from ROCKET AF. Cardiol Ther. 2019 Dec;8(2):283-295. doi: 10.1007/s40119-019-00146-6. Epub 2019 Aug 2. PMID 31376090
- [Derived] Quinn GR, Hellkamp AS, Hankey GJ, Becker RC, Berkowitz SD, Breithardt G, Fava M, Fox KAA, Halperin JL, Mahaffey KW, Nessel CC, Patel MR, Piccini JP, Singer DE. Selective Serotonin Reuptake Inhibitors and Bleeding Risk in Anticoagulated Patients With Atrial Fibrillation: An Analysis From the ROCKET AF Trial. J Am Heart Assoc. 2018 Aug 7;7(15):e008755. doi: 10.1161/JAHA.118.008755. PMID 30371223
- [Derived] Chen ST, Hellkamp AS, Becker RC, Berkowitz SD, Breithardt G, Fox KAA, Hacke W, Halperin JL, Hankey GJ, Mahaffey KW, Nessel CC, Piccini JP, Singer DE, Patel MR, Melloni C. Efficacy and safety of rivaroxaban vs. warfarin in patients with non-valvular atrial fibrillation and a history of cancer: observations from ROCKET AF. Eur Heart J Qual Care Clin Outcomes. 2019 Apr 1;5(2):145-152. doi: 10.1093/ehjqcco/qcy040. PMID 30219887
- [Derived] Chen ST, Hellkamp AS, Becker RC, Berkowitz SD, Breithardt G, Fox KAA, Hacke W, Halperin JL, Hankey GJ, Mahaffey KW, Nessel CC, Piccini JP, Singer DE, Patel MR. Impact of polyvascular disease on patients with atrial fibrillation: Insights from ROCKET AF. Am Heart J. 2018 Jun;200:102-109. doi: 10.1016/j.ahj.2018.02.013. Epub 2018 Feb 27. PMID 29898836
- [Derived] Leef GC, Hellkamp AS, Patel MR, Becker RC, Berkowitz SD, Breithardt G, Halperin JL, Hankey GJ, Hacke W, Nessel CC, Singer DE, Fox KAA, Mahaffey KW, Piccini JP. Safety and Efficacy of Rivaroxaban in Patients With Cardiac Implantable Electronic Devices: Observations From the ROCKET AF Trial. J Am Heart Assoc. 2017 Jun 14;6(6):e004663. doi: 10.1161/JAHA.116.004663. PMID 28615214
- [Derived] Balla SR, Cyr DD, Lokhnygina Y, Becker RC, Berkowitz SD, Breithardt G, Fox KAA, Hacke W, Halperin JL, Hankey GJ, Mahaffey KW, Nessel CC, Piccini JP, Singer DE, Patel MR. Relation of Risk of Stroke in Patients With Atrial Fibrillation to Body Mass Index (from Patients Treated With Rivaroxaban and Warfarin in the Rivaroxaban Once Daily Oral Direct Factor Xa Inhibition Compared with Vitamin K Antagonism for Prevention of Stroke and Embolism Trial in Atrial Fibrillation Trial). Am J Cardiol. 2017 Jun 15;119(12):1989-1996. doi: 10.1016/j.amjcard.2017.03.028. Epub 2017 Mar 29. PMID 28477860
- [Derived] Sun Y, Hu D, Stevens S, Lokhnygina Y, Becker RC, Berkowitz SD, Breithardt G, Hacke W, Halperin JL, Hankey GJ, Mahaffey KW, Nessel CC, Piccini JP, Singer DE, Fox KAA, Patel MR. Efficacy and safety of rivaroxaban versus warfarin in patients from mainland China with nonvalvular atrial fibrillation: A subgroup analysis from the ROCKET AF trial. Thromb Res. 2017 Aug;156:184-190. doi: 10.1016/j.thromres.2017.04.010. Epub 2017 Apr 13. PMID 28433206
- [Derived] Lindner SM, Fordyce CB, Hellkamp AS, Lokhnygina Y, Piccini JP, Breithardt G, Mahaffey KW, Singer DE, Hacke W, Halperin JL, Hankey GJ, Berkowitz SD, Nessel CC, Becker RC, Fox KA, Patel MR; ROCKET AF Steering Committee and Investigators. Treatment Consistency Across Levels of Baseline Renal Function With Rivaroxaban or Warfarin: A ROCKET AF (Rivaroxaban Once-Daily, Oral, Direct Factor Xa Inhibition Compared With Vitamin K Antagonism for Prevention of Stroke and Embolism Trial in Atrial Fibrillation) Analysis. Circulation. 2017 Mar 7;135(10):1001-1003. doi: 10.1161/CIRCULATIONAHA.116.024666. No abstract available. PMID 28264892
- [Derived] Fordyce CB, Hellkamp AS, Lokhnygina Y, Lindner SM, Piccini JP, Becker RC, Berkowitz SD, Breithardt G, Fox KA, Mahaffey KW, Nessel CC, Singer DE, Patel MR; ROCKET AF Steering Committee and Investigators. On-Treatment Outcomes in Patients With Worsening Renal Function With Rivaroxaban Compared With Warfarin: Insights From ROCKET AF. Circulation. 2016 Jul 5;134(1):37-47. doi: 10.1161/CIRCULATIONAHA.116.021890. PMID 27358435
- [Derived] Pokorney SD, Piccini JP, Stevens SR, Patel MR, Pieper KS, Halperin JL, Breithardt G, Singer DE, Hankey GJ, Hacke W, Becker RC, Berkowitz SD, Nessel CC, Mahaffey KW, Fox KA, Califf RM; ROCKET AF Steering Committee & Investigators; ROCKET AF Steering Committee Investigators. Cause of Death and Predictors of All-Cause Mortality in Anticoagulated Patients With Nonvalvular Atrial Fibrillation: Data From ROCKET AF. J Am Heart Assoc. 2016 Mar 8;5(3):e002197. doi: 10.1161/JAHA.115.002197. PMID 26955859
- [Derived] Breithardt G, Baumgartner H, Berkowitz SD, Hellkamp AS, Piccini JP, Lokhnygina Y, Halperin JL, Singer DE, Hankey GJ, Hacke W, Becker RC, Nessel CC, Mahaffey KW, Califf RM, Fox KA, Patel MR; ROCKET AF Steering Committee & Investigators. Native valve disease in patients with non-valvular atrial fibrillation on warfarin or rivaroxaban. Heart. 2016 Jul 1;102(13):1036-43. doi: 10.1136/heartjnl-2015-308120. Epub 2016 Feb 17. PMID 26888572
- [Derived] Piccini JP, Hellkamp AS, Washam JB, Becker RC, Breithardt G, Berkowitz SD, Halperin JL, Hankey GJ, Hacke W, Mahaffey KW, Nessel CC, Singer DE, Fox KA, Patel MR. Polypharmacy and the Efficacy and Safety of Rivaroxaban Versus Warfarin in the Prevention of Stroke in Patients With Nonvalvular Atrial Fibrillation. Circulation. 2016 Jan 26;133(4):352-60. doi: 10.1161/CIRCULATIONAHA.115.018544. Epub 2015 Dec 16. PMID 26673560
- [Derived] Bansilal S, Bloomgarden Z, Halperin JL, Hellkamp AS, Lokhnygina Y, Patel MR, Becker RC, Breithardt G, Hacke W, Hankey GJ, Nessel CC, Singer DE, Berkowitz SD, Piccini JP, Mahaffey KW, Fox KA; ROCKET AF Steering Committee and Investigators. Efficacy and safety of rivaroxaban in patients with diabetes and nonvalvular atrial fibrillation: the Rivaroxaban Once-daily, Oral, Direct Factor Xa Inhibition Compared with Vitamin K Antagonism for Prevention of Stroke and Embolism Trial in Atrial Fibrillation (ROCKET AF Trial). Am Heart J. 2015 Oct;170(4):675-682.e8. doi: 10.1016/j.ahj.2015.07.006. Epub 2015 Jul 17. PMID 26386791
- [Derived] Washam JB, Stevens SR, Lokhnygina Y, Halperin JL, Breithardt G, Singer DE, Mahaffey KW, Hankey GJ, Berkowitz SD, Nessel CC, Fox KA, Califf RM, Piccini JP, Patel MR; ROCKET AF Steering Committee and Investigators. Digoxin use in patients with atrial fibrillation and adverse cardiovascular outcomes: a retrospective analysis of the Rivaroxaban Once Daily Oral Direct Factor Xa Inhibition Compared with Vitamin K Antagonism for Prevention of Stroke and Embolism Trial in Atrial Fibrillation (ROCKET AF). Lancet. 2015 Jun 13;385(9985):2363-70. doi: 10.1016/S0140-6736(14)61836-5. Epub 2015 Mar 6. PMID 25749644
- [Derived] Singer DE, Hellkamp AS, Yuan Z, Lokhnygina Y, Patel MR, Piccini JP, Hankey GJ, Breithardt G, Halperin JL, Becker RC, Hacke W, Nessel CC, Mahaffey KW, Fox KA, Califf RM; ROCKET AF Investigators. Alternative calculations of individual patient time in therapeutic range while taking warfarin: results from the ROCKET AF trial. J Am Heart Assoc. 2015 Mar 3;4(3):e001349. doi: 10.1161/JAHA.114.001349. PMID 25736441
- [Derived] Girgis IG, Patel MR, Peters GR, Moore KT, Mahaffey KW, Nessel CC, Halperin JL, Califf RM, Fox KA, Becker RC. Population pharmacokinetics and pharmacodynamics of rivaroxaban in patients with non-valvular atrial fibrillation: results from ROCKET AF. J Clin Pharmacol. 2014 Aug;54(8):917-27. doi: 10.1002/jcph.288. Epub 2014 Mar 26. PMID 24668660
- [Derived] Sherwood MW, Douketis JD, Patel MR, Piccini JP, Hellkamp AS, Lokhnygina Y, Spyropoulos AC, Hankey GJ, Singer DE, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Becker RC; ROCKET AF Investigators. Outcomes of temporary interruption of rivaroxaban compared with warfarin in patients with nonvalvular atrial fibrillation: results from the rivaroxaban once daily, oral, direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and embolism trial in atrial fibrillation (ROCKET AF). Circulation. 2014 May 6;129(18):1850-9. doi: 10.1161/CIRCULATIONAHA.113.005754. Epub 2014 Feb 19. PMID 24552831
- [Derived] Goodman SG, Wojdyla DM, Piccini JP, White HD, Paolini JF, Nessel CC, Berkowitz SD, Mahaffey KW, Patel MR, Sherwood MW, Becker RC, Halperin JL, Hacke W, Singer DE, Hankey GJ, Breithardt G, Fox KA, Califf RM; ROCKET AF Investigators. Factors associated with major bleeding events: insights from the ROCKET AF trial (rivaroxaban once-daily oral direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and embolism trial in atrial fibrillation). J Am Coll Cardiol. 2014 Mar 11;63(9):891-900. doi: 10.1016/j.jacc.2013.11.013. Epub 2013 Dec 4. PMID 24315894
- [Derived] Mahaffey KW, Wojdyla D, Hankey GJ, White HD, Nessel CC, Piccini JP, Patel MR, Berkowitz SD, Becker RC, Halperin JL, Singer DE, Califf RM, Fox KA, Breithardt G, Hacke W. Clinical outcomes with rivaroxaban in patients transitioned from vitamin K antagonist therapy: a subgroup analysis of a randomized trial. Ann Intern Med. 2013 Jun 18;158(12):861-8. doi: 10.7326/0003-4819-158-12-201306180-00003. PMID 23778903
- [Derived] van Diepen S, Hellkamp AS, Patel MR, Becker RC, Breithardt G, Hacke W, Halperin JL, Hankey GJ, Nessel CC, Singer DE, Berkowitz SD, Califf RM, Fox KA, Mahaffey KW. Efficacy and safety of rivaroxaban in patients with heart failure and nonvalvular atrial fibrillation: insights from ROCKET AF. Circ Heart Fail. 2013 Jul;6(4):740-7. doi: 10.1161/CIRCHEARTFAILURE.113.000212. Epub 2013 May 30. PMID 23723250
- [Derived] Singer DE, Hellkamp AS, Piccini JP, Mahaffey KW, Lokhnygina Y, Pan G, Halperin JL, Becker RC, Breithardt G, Hankey GJ, Hacke W, Nessel CC, Patel MR, Califf RM, Fox KA; ROCKET AF Investigators. Impact of global geographic region on time in therapeutic range on warfarin anticoagulant therapy: data from the ROCKET AF clinical trial. J Am Heart Assoc. 2013 Feb 19;2(1):e000067. doi: 10.1161/JAHA.112.000067. PMID 23525418
- [Derived] Piccini JP, Stevens SR, Lokhnygina Y, Patel MR, Halperin JL, Singer DE, Hankey GJ, Hacke W, Becker RC, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Breithardt G; ROCKET AF Steering Committee & Investigators. Outcomes after cardioversion and atrial fibrillation ablation in patients treated with rivaroxaban and warfarin in the ROCKET AF trial. J Am Coll Cardiol. 2013 May 14;61(19):1998-2006. doi: 10.1016/j.jacc.2013.02.025. Epub 2013 Mar 14. PMID 23500298
- [Derived] Piccini JP, Stevens SR, Chang Y, Singer DE, Lokhnygina Y, Go AS, Patel MR, Mahaffey KW, Halperin JL, Breithardt G, Hankey GJ, Hacke W, Becker RC, Nessel CC, Fox KA, Califf RM; ROCKET AF Steering Committee and Investigators. Renal dysfunction as a predictor of stroke and systemic embolism in patients with nonvalvular atrial fibrillation: validation of the R(2)CHADS(2) index in the ROCKET AF (Rivaroxaban Once-daily, oral, direct factor Xa inhibition Compared with vitamin K antagonism for prevention of stroke and Embolism Trial in Atrial Fibrillation) and ATRIA (AnTicoagulation and Risk factors In Atrial fibrillation) study cohorts. Circulation. 2013 Jan 15;127(2):224-32. doi: 10.1161/CIRCULATIONAHA.112.107128. Epub 2012 Dec 3. PMID 23212720
- [Derived] Hankey GJ, Patel MR, Stevens SR, Becker RC, Breithardt G, Carolei A, Diener HC, Donnan GA, Halperin JL, Mahaffey KW, Mas JL, Massaro A, Norrving B, Nessel CC, Paolini JF, Roine RO, Singer DE, Wong L, Califf RM, Fox KA, Hacke W; ROCKET AF Steering Committee Investigators. Rivaroxaban compared with warfarin in patients with atrial fibrillation and previous stroke or transient ischaemic attack: a subgroup analysis of ROCKET AF. Lancet Neurol. 2012 Apr;11(4):315-22. doi: 10.1016/S1474-4422(12)70042-X. Epub 2012 Mar 7. PMID 22402056
- [Derived] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Derived] ROCKET AF Study Investigators. Rivaroxaban-once daily, oral, direct factor Xa inhibition compared with vitamin K antagonism for prevention of stroke and Embolism Trial in Atrial Fibrillation: rationale and design of the ROCKET AF study. Am Heart J. 2010 Mar;159(3):340-347.e1. doi: 10.1016/j.ahj.2009.11.025. PMID 20211293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study, an efficacy and safety study of Rivaroxaban with Warfarin for the prevention of stroke and non-central nervous system systemic embolism in patients with non-valvular atrial fibrillation, was conducted from 18 December 2006 to 07 September 2010. Patients were recruited at 1,170 study centers located in 45 countries worldwide.
Pre-assignment Details: A total of 14,269 patients were randomized in the study. Five patients were randomized twice bringing the number of randomized unique patients to 14,264. A total of 14,236 (7111 and 7125 patients in the rivaroxaban and warfarin groups, respectively) unique patients took at least 1 dose of study medication and were included in the Safety Population.
Groups:
- Rivaroxaban: Rivaroxaban 15 mg p.o. once daily or Rivaroxaban 20 mg p.o. once daily
- Warfarin: Warfarin (1 mg, 2.5 mg, or 5 mg p.o. once daily)
Period: Overall Study
Arm/Group | Rivaroxaban | Warfarin
Started | 7111 | 7125
Completed | 4591 | 4657
Not Completed | 2520 | 2468
Not completed — Adverse Event | 993 | 919
Not completed — Non-compliant with study medication | 134 | 164
Not completed — Consent withdrawn | 671 | 673
Not completed — Investigator dec./not protocol-related | 191 | 178
Not completed — Lost to Follow-up | 6 | 8
Not completed — Protocol Violation | 142 | 124
Not completed — Clinical efficacy endpoint reached | 300 | 332
Not completed — Study terminated by sponsor | 82 | 69
Not completed — Missing/incomplete data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban | Warfarin | Total
Number analyzed (Participants) | 7111 | 7125 | 14236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1646 | 1642 | 3288
  >=65 years | 5465 | 5483 | 10948
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age Continuous | 71.2 (9.45) | 71.2 (9.39) | 71.2 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2819 | 2826 | 5645
  Male | 4292 | 4299 | 8591
Region of Enrollment [Number; unit: participants]
  Argentina | 284 | 285 | 569
  Australia | 120 | 122 | 242
  Austria | 16 | 16 | 32
  Belgium | 49 | 47 | 96
  Brazil | 241 | 242 | 483
  Bulgaria | 337 | 339 | 676
  Canada | 372 | 375 | 747
  Chile | 144 | 142 | 286
  China | 249 | 246 | 495
  Colombia | 134 | 133 | 267
  Czech Republic | 299 | 299 | 598
  Denmark | 60 | 61 | 121
  Finland | 9 | 7 | 16
  France | 35 | 36 | 71
  Germany | 263 | 265 | 528
  Greece | 15 | 14 | 29
  Hungary | 119 | 118 | 237
  India | 133 | 135 | 268
  Israel | 94 | 94 | 188
  Italy | 69 | 69 | 138
  Korea (South) | 103 | 100 | 203
  Lithuania | 122 | 122 | 244
  Malaysia | 26 | 25 | 51
  Mexico | 83 | 85 | 168
  Netherlands | 80 | 81 | 161
  New Zealand | 58 | 58 | 116
  Norway | 25 | 24 | 49
  Peru | 42 | 42 | 84
  Philippines | 185 | 183 | 368
  Poland | 263 | 264 | 527
  Romania | 391 | 391 | 782
  Russia | 645 | 645 | 1290
  Singapore | 21 | 23 | 44
  South Africa | 122 | 125 | 247
  Spain | 124 | 124 | 248
  Sweden | 12 | 16 | 28
  Switzerland | 3 | 4 | 7
  Taiwan | 78 | 79 | 157
  Thailand | 43 | 44 | 87
  Turkey | 50 | 51 | 101
  Ukraine | 505 | 504 | 1009
  United Kingdom | 79 | 80 | 159
  United States | 962 | 964 | 1926
  Venezuela | 11 | 9 | 20
  Hong Kong | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: The Composite Event of Stroke/Non-CNS Systemic Embolism: Primary Efficacy (Non-Inferiority)
Description: The number of patients with the first occurrence of a stroke or non-CNS systemic embolism while on treatment (defined as the time interval from the first dose to the last dose of study drug plus 2 days). The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: The per-protocol (PP) population consisted of all randomized unique patients excluding those who had specific pre-defined major protocol deviations that occurred by the time of enrollment into the study or during the trial. Site 042012 with GCP violation was excluded.
Measure: Number; unit: Patients
Groups:
- Rivaroxaban: Rivaroxaban 20 mg p.o. once daily or matching placebo (15 mg p.o. once daily for patients with a calculated creatinine clearance of 30 - 49 mL/min. at baseline)
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 6958 | 7004
Patients | 188 | 241
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Test type: Non-Inferiority or Equivalence — Alternative hypothesis of non-inferiority (NI) by a NI margin of 1.46 in hazard ratio (HR) based on on-treatment data from the per protocol population. The required number of primary efficacy endpoint events was determined based on the following assumptions: NI margin of 1.46, 1-sided alpha of 0.025, power of >95% when true HR is 1, and exponential distributions. The margin was selected based on clinical appropriateness and quantitative analysis of relevant studies in Hart et al; p < 0.001, Cox Proportional Hazards model — The p-value is not adjusted for multiple comparisons. The alpha threshold for statistical significance is 0.025 (1-sided); (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.66 to 0.96]

2. Primary Outcome: The Composite of Event of Stroke/Non-CNS Systemic Embolism: Primary Efficacy (Superiority)
Description: as for outcome 1
Time Frame: Up to 4 years
Population: The safety population consisted of all randomized unique patients who took at least 1 dose of study medication after randomization during the double-blind treatment period. Site 042012 with GCP violation was excluded.
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 189 | 243
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.015, Cox Proportional Hazards model — The p-value Is not adjusted for multiple comparisons. The alpha threshold for statistical significance is 0.05 (2-sided); (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.95]

3. Primary Outcome: The Composite Event of Major/Non-major Clinically Relevant Bleeding Events: Primary Safety
Description: The number of patients with the first occurrence of a major or non-major clinically relevant bleeding event while on treatment. The statistical analysis is based on time from the first dose of study drug to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: The safety population consisted of all randomized unique patients who took at least 1 dose of study medication after randomization during the double-blind treatment period.
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7111 | 7125
Patients | 1475 | 1449
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternate hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.442, Cox Proportional Hazards model — The p-value is not adjusted for mulitple comparisons. The alpha threshold for statistical significance is 0.05 (2-sided); (non-stratified) Cox Proportional Hazards model with treatment as a covariate; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.96 to 1.11]

4. Secondary Outcome: The Composite Event of Stroke/Non-CNS Systemic Embolism/Vascular Death
Description: The number of patients with the first occurrence of a stroke, non-CNS systemic embolism, or vascular death while on treatment. The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7125
Patients | 346 | 410
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.034, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 0.99]

5. Secondary Outcome: The Composite Event of Stroke/Non-CNS Systemic Embolism/Myocardial Infarction/Vascular Death
Description: The number of patients with the first occurrence of a stroke, non-CNS systemic embolism, myocardial infarction, or vascular death while on treatment. The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 433 | 519
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.010, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.74 to 0.96]

6. Secondary Outcome: The Individual Components of the Composite Primary and Major Secondary Efficacy Outcome Measures: Stroke
Description: The number of patients with the first occurrence of a stroke while on treatment. The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 184 | 221
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.092, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as a covariate; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.03]

7. Secondary Outcome: The Individual Components of the Composite Primary and Major Secondary Efficacy Outcome Measures: Non-CNS Systemic Embolism
Description: The number of patients with the first occurrence of a non-CNS systemic embolism while on treatment. The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 5 | 22
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.003, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.09 to 0.61]

8. Secondary Outcome: The Individual Components of the Composite Primary and Major Secondary Efficacy Outcome Measures: Myocardial Infarction
Description: The number of patients with the first occurrence of a myocardial infarction while on treatment. The statistical analysis is based on time from randomization to the first occurrence of the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 101 | 126
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.121, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as a covariate; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.63 to 1.06]

9. Secondary Outcome: The Individual Components of the Composite Primary and Major Secondary Efficacy Outcome Measures: Vascular Death
Description: The number of patients with the occurrence of vascular death while on treatment. The statistical analysis is based on time from randomization to the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7082
Patients | 170 | 193
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.289, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as a covariate; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.73 to 1.10]

10. Secondary Outcome: All-cause Mortality
Description: The number of patients who died due to any cause while on treatment. The statistical analysis is based on time from randomization to the event while on treatment.
Time Frame: Up to 4 years
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Rivaroxaban | Warfarin
Number analyzed (Participants) | 7061 | 7125
Patients | 208 | 250
Statistical Analysis 1: Comparison: Rivaroxaban vs Warfarin; Alternative hypothesis of superiority based on on-treatment data from the safety population; Test type: Superiority or Other; p = 0.073, Cox Proportional Hazards model — [p-value comment as in outcome 2, analysis 1]; (non-stratified) Cox Proportional Hazards model with treatment as covariate; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.02]

ADVERSE EVENTS:
Arm/Group | Rivaroxaban | Warfarin
Serious Adverse Events (participants affected / at risk) | 2649/7111 | 2720/7125
Other Adverse Events (participants affected / at risk) | 2537/7111 | 2573/7125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=7111) | Warfarin (N=7125)
Anaemia (Blood and lymphatic system disorders) | 68 | 31
Anaemia Haemolytic Autoimmune (Blood and lymphatic system disorders) | 1 | 0
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 0 | 2
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 5 | 5
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypocoagulable State (Blood and lymphatic system disorders) | 0 | 1
Hypoplastic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 16 | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 2 | 0
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 3 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic Infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 5 | 8
Acute Left Ventricular Failure (Cardiac disorders) | 5 | 4
Acute Myocardial Infarction (Cardiac disorders) | 6 | 11
Acute Right Ventricular Failure (Cardiac disorders) | 0 | 1
Adams-Stokes Syndrome (Cardiac disorders) | 0 | 2
Angina Pectoris (Cardiac disorders) | 31 | 33
Angina Unstable (Cardiac disorders) | 74 | 92
Aortic Valve Disease (Cardiac disorders) | 0 | 1
Aortic Valve Disease Mixed (Cardiac disorders) | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 1 | 1
Aortic Valve Stenosis (Cardiac disorders) | 4 | 8
Arrhythmia (Cardiac disorders) | 9 | 6
Arteriosclerosis Coronary Artery (Cardiac disorders) | 7 | 3
Atrial Fibrillation (Cardiac disorders) | 158 | 161
Atrial Flutter (Cardiac disorders) | 10 | 17
Atrial Tachycardia (Cardiac disorders) | 0 | 1
Atrial Thrombosis (Cardiac disorders) | 2 | 3
Atrioventricular Block (Cardiac disorders) | 2 | 4
Atrioventricular Block Complete (Cardiac disorders) | 12 | 9
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 2
Bradyarrhythmia (Cardiac disorders) | 3 | 3
Bradycardia (Cardiac disorders) | 35 | 23
Cardiac Amyloidosis (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 15 | 33
Cardiac Asthma (Cardiac disorders) | 3 | 1
Cardiac Disorder (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 283 | 309
Cardiac Failure Acute (Cardiac disorders) | 40 | 36
Cardiac Failure Chronic (Cardiac disorders) | 26 | 43
Cardiac Failure Congestive (Cardiac disorders) | 178 | 206
Cardiac Tamponade (Cardiac disorders) | 1 | 2
Cardiac Valve Disease (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 7 | 10
Cardiogenic Shock (Cardiac disorders) | 14 | 10
Cardiomyopathy (Cardiac disorders) | 3 | 6
Cardiopulmonary Failure (Cardiac disorders) | 2 | 1
Cardiovascular Insufficiency (Cardiac disorders) | 1 | 2
Congestive Cardiomyopathy (Cardiac disorders) | 3 | 1
Cor Pulmonale (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 29 | 33
Coronary Artery Insufficiency (Cardiac disorders) | 1 | 3
Coronary Artery Stenosis (Cardiac disorders) | 1 | 3
Electromechanical Dissociation (Cardiac disorders) | 3 | 1
Heart Valve Stenosis (Cardiac disorders) | 0 | 1
Hypertensive Heart Disease (Cardiac disorders) | 3 | 0
Hypertrophic Cardiomyopathy (Cardiac disorders) | 0 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 | 3
Left Ventricular Dysfunction (Cardiac disorders) | 3 | 2
Left Ventricular Failure (Cardiac disorders) | 11 | 12
Mitral Valve Incompetence (Cardiac disorders) | 7 | 6
Myocardial Infarction (Cardiac disorders) | 19 | 22
Myocardial Ischaemia (Cardiac disorders) | 6 | 6
Myocarditis (Cardiac disorders) | 0 | 1
Nodal Arrhythmia (Cardiac disorders) | 0 | 2
Nodal Rhythm (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 3
Pericardial Effusion (Cardiac disorders) | 4 | 1
Pericardial Haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 4 | 2
Sick Sinus Syndrome (Cardiac disorders) | 37 | 25
Sinus Arrest (Cardiac disorders) | 3 | 1
Sinus Arrhythmia (Cardiac disorders) | 4 | 4
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 10 | 3
Tachycardia (Cardiac disorders) | 6 | 8
Tachycardia Paroxysmal (Cardiac disorders) | 0 | 1
Torsade De Pointes (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 4
Ventricular Asystole (Cardiac disorders) | 0 | 1
Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 1 | 3
Ventricular Fibrillation (Cardiac disorders) | 18 | 13
Ventricular Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 16 | 19
Gastrointestinal Angiodysplasia Haemorrhagic (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 3 | 4
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 | 0
Ear Haemorrhage (Ear and labyrinth disorders) | 2 | 0
External Ear Inflammation (Ear and labyrinth disorders) | 0 | 1
Inner Ear Disorder (Ear and labyrinth disorders) | 0 | 1
Meniere's Disease (Ear and labyrinth disorders) | 1 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 2 | 2
Vertigo (Ear and labyrinth disorders) | 10 | 10
Vertigo Positional (Ear and labyrinth disorders) | 1 | 1
Vestibular Disorder (Ear and labyrinth disorders) | 2 | 2
Cushing's Syndrome (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 6 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Primary Hyperaldosteronism (Endocrine disorders) | 1 | 0
Amaurosis Fugax (Eye disorders) | 1 | 0
Angle Closure Glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 13 | 31
Cataract Diabetic (Eye disorders) | 0 | 1
Chorioretinal Atrophy (Eye disorders) | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 1 | 3
Dacryostenosis Acquired (Eye disorders) | 1 | 0
Diabetic Retinopathy (Eye disorders) | 1 | 0
Eye Haemorrhage (Eye disorders) | 4 | 2
Glaucoma (Eye disorders) | 4 | 2
Glaucomatocyclitic Crises (Eye disorders) | 1 | 0
Hyphaema (Eye disorders) | 0 | 1
Keratopathy (Eye disorders) | 0 | 1
Macular Degeneration (Eye disorders) | 0 | 1
Macular Hole (Eye disorders) | 0 | 1
Macular Oedema (Eye disorders) | 1 | 0
Open Angle Glaucoma (Eye disorders) | 1 | 0
Retinal Artery Thrombosis (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 2 | 5
Retinal Haemorrhage (Eye disorders) | 2 | 3
Retinal Vein Occlusion (Eye disorders) | 1 | 1
Retinal Vein Thrombosis (Eye disorders) | 1 | 1
Retinopathy Haemorrhagic (Eye disorders) | 0 | 1
Retinoschisis (Eye disorders) | 0 | 1
Scleral Haemorrhage (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Ulcerative Keratitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Vitreous Degeneration (Eye disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 3 | 1
Abdominal Adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 2
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 | 2
Abdominal Mass (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 10 | 5
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 2
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 | 4
Acute Abdomen (Gastrointestinal disorders) | 1 | 2
Anal Fistula (Gastrointestinal disorders) | 1 | 2
Anal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 2 | 4
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic Obstruction (Gastrointestinal disorders) | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 9 | 8
Constipation (Gastrointestinal disorders) | 8 | 6
Dental Caries (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 9
Diverticular Perforation (Gastrointestinal disorders) | 1 | 3
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 4
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 3
Duodenal Polyp (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 4 | 3
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 4 | 4
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 2
Enterocolitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Femoral Hernia, Obstructive (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 9 | 7
Gastric Polyps (Gastrointestinal disorders) | 4 | 0
Gastric Ulcer (Gastrointestinal disorders) | 2 | 4
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 11 | 9
Gastric Varices (Gastrointestinal disorders) | 0 | 1
Gastric Varices Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 10 | 4
Gastritis Erosive (Gastrointestinal disorders) | 2 | 9
Gastritis Haemorrhagic (Gastrointestinal disorders) | 7 | 1
Gastroduodenal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroduodenal Ulcer (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 88 | 62
Gastrointestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 4
Gastrooesophagitis (Gastrointestinal disorders) | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 5 | 3
Haematemesis (Gastrointestinal disorders) | 3 | 4
Haematochezia (Gastrointestinal disorders) | 3 | 4
Haemorrhagic Erosive Gastritis (Gastrointestinal disorders) | 4 | 5
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 6 | 4
Haemorrhoids (Gastrointestinal disorders) | 7 | 4
Hiatus Hernia (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 5 | 4
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 29 | 21
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 | 1
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 3 | 0
Intestinal Cyst (Gastrointestinal disorders) | 0 | 1
Intestinal Dilatation (Gastrointestinal disorders) | 0 | 1
Intestinal Haemorrhage (Gastrointestinal disorders) | 4 | 4
Intestinal Infarction (Gastrointestinal disorders) | 2 | 3
Intestinal Ischaemia (Gastrointestinal disorders) | 2 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 4 | 6
Intestinal Perforation (Gastrointestinal disorders) | 1 | 1
Intestinal Polyp (Gastrointestinal disorders) | 2 | 1
Intestinal Strangulation (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 | 1
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 2 | 2
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 19 | 15
Lumbar Hernia (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 2 | 0
Mechanical Ileus (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 29 | 18
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 0 | 2
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 3 | 2
Oesophageal Disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Oesophageal Rupture (Gastrointestinal disorders) | 1 | 0
Oesophageal Spasm (Gastrointestinal disorders) | 1 | 0
Oesophageal Stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 1
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophagitis Haemorrhagic (Gastrointestinal disorders) | 1 | 1
Pancreatic Cyst (Gastrointestinal disorders) | 0 | 1
Pancreatic Mass (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 6 | 2
Pancreatitis Acute (Gastrointestinal disorders) | 7 | 6
Pancreatitis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Pancreatitis Relapsing (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 2 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 3 | 4
Peritoneal Necrosis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 24 | 26
Rectal Polyp (Gastrointestinal disorders) | 1 | 2
Rectal Ulcer (Gastrointestinal disorders) | 1 | 0
Rectal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Regurgitation (Gastrointestinal disorders) | 0 | 1
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 2
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 4
Subileus (Gastrointestinal disorders) | 1 | 2
Tongue Haemorrhage (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 3
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 53 | 34
Varices Oesophageal (Gastrointestinal disorders) | 1 | 1
Volvulus (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 4 | 3
Cardiac Death (General disorders) | 0 | 2
Catheter Site Haemorrhage (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 0 | 4
Chest Pain (General disorders) | 37 | 44
Chills (General disorders) | 1 | 0
Death (General disorders) | 19 | 23
Device Capturing Issue (General disorders) | 1 | 0
Device Dislocation (General disorders) | 2 | 1
Device Lead Damage (General disorders) | 1 | 0
Device Malfunction (General disorders) | 6 | 5
Device Occlusion (General disorders) | 4 | 0
Device Power Source Issue (General disorders) | 1 | 1
Gait Disturbance (General disorders) | 1 | 1
General Physical Health Deterioration (General disorders) | 0 | 3
Generalised Oedema (General disorders) | 3 | 1
Hernia (General disorders) | 0 | 2
Hernia Pain (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Impaired Healing (General disorders) | 1 | 1
Implant Site Haemorrhage (General disorders) | 0 | 1
Implant Site Reaction (General disorders) | 0 | 1
Injury Associated with Device (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 3
Medical Device Complication (General disorders) | 2 | 1
Multi-Organ Failure (General disorders) | 10 | 6
Non-Cardiac Chest Pain (General disorders) | 15 | 16
Oedema (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 5 | 4
Pelvic Mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 6
Sudden Cardiac Death (General disorders) | 12 | 13
Sudden Death (General disorders) | 80 | 68
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Thrombosis in Device (General disorders) | 0 | 1
Vessel Puncture Site Haemorrhage (General disorders) | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 2 | 1
Bile Duct Stone (Hepatobiliary disorders) | 5 | 7
Biliary Colic (Hepatobiliary disorders) | 2 | 2
Cardiac Cirrhosis (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 7 | 2
Cholangitis Acute (Hepatobiliary disorders) | 1 | 0
Cholangitis Sclerosing (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 9 | 13
Cholecystitis Acute (Hepatobiliary disorders) | 23 | 15
Cholecystitis Chronic (Hepatobiliary disorders) | 6 | 0
Cholelithiasis (Hepatobiliary disorders) | 20 | 16
Cholelithiasis Obstructive (Hepatobiliary disorders) | 0 | 1
Cryptogenic Cirrhosis (Hepatobiliary disorders) | 0 | 2
Cytolytic Hepatitis (Hepatobiliary disorders) | 2 | 0
Gallbladder Fistula (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 3 | 2
Hepatic Congestion (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 2 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 1
Hepatitis Acute (Hepatobiliary disorders) | 1 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 | 3
Jaundice (Hepatobiliary disorders) | 0 | 2
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 2
Jaundice Hepatocellular (Hepatobiliary disorders) | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Anaphylactic Shock (Immune system disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 2 | 1
Hypersensitivity (Immune system disorders) | 3 | 0
Skin Graft Rejection (Immune system disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 2 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 1
Abscess Neck (Infections and infestations) | 1 | 0
Abscess of External Auditory Meatus (Infections and infestations) | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0
Amoebic Dysentery (Infections and infestations) | 1 | 0
Anal Abscess (Infections and infestations) | 3 | 0
Appendiceal Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 12 | 7
Appendicitis Perforated (Infections and infestations) | 2 | 1
Arthritis Bacterial (Infections and infestations) | 2 | 1
Arthritis Infective (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 2 | 2
Bacterial Infection (Infections and infestations) | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0
Blister Infected (Infections and infestations) | 1 | 0
Breast Cellulitis (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 38 | 32
Bronchitis Bacterial (Infections and infestations) | 1 | 1
Bronchitis Viral (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 11 | 12
Bursitis Infective Staphylococcal (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 42 | 64
Cellulitis Pharyngeal (Infections and infestations) | 1 | 0
Cellulitis of Male External Genital Organ (Infections and infestations) | 1 | 0
Cervicitis (Infections and infestations) | 0 | 1
Cholecystitis Infective (Infections and infestations) | 2 | 1
Clostridial Infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 2 | 1
Dengue Fever (Infections and infestations) | 0 | 4
Device Related Infection (Infections and infestations) | 3 | 1
Diabetic Foot Infection (Infections and infestations) | 2 | 0
Diabetic Gangrene (Infections and infestations) | 0 | 2
Diarrhoea Infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 7 | 10
Ear Infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Encephalitis Herpes (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 3 | 0
Endocarditis Bacterial (Infections and infestations) | 1 | 0
Enterococcal Bacteraemia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 17 | 15
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Extradural Abscess (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 4 | 5
Gastroenteritis (Infections and infestations) | 18 | 38
Gastroenteritis Norovirus (Infections and infestations) | 1 | 1
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Groin Abscess (Infections and infestations) | 0 | 1
Haematoma Infection (Infections and infestations) | 1 | 1
Helicobacter Gastritis (Infections and infestations) | 2 | 1
Hepatitis B (Infections and infestations) | 1 | 2
Hepatitis C (Infections and infestations) | 3 | 5
Hepatitis E (Infections and infestations) | 1 | 0
Hepatitis Viral (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 6 | 6
Herpes Zoster Ophthalmic (Infections and infestations) | 0 | 1
Herpes Zoster Oticus (Infections and infestations) | 1 | 0
Implant Site Infection (Infections and infestations) | 3 | 2
Incision Site Abscess (Infections and infestations) | 1 | 0
Infected Epidermal Cyst (Infections and infestations) | 0 | 1
Infected Sebaceous Cyst (Infections and infestations) | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 3 | 1
Infection (Infections and infestations) | 2 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 5 | 3
Infusion Site Infection (Infections and infestations) | 1 | 0
Intertrigo Candida (Infections and infestations) | 0 | 1
Intervertebral Discitis (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 2
Labyrinthitis (Infections and infestations) | 2 | 1
Laryngitis Bacterial (Infections and infestations) | 0 | 1
Leptospirosis (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 16 | 13
Localised Infection (Infections and infestations) | 3 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 4 | 4
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 13 | 7
Lung Infection Pseudomonal (Infections and infestations) | 1 | 0
Lyme Disease (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Meningitis Bacterial (Infections and infestations) | 1 | 0
Meningitis Pneumococcal (Infections and infestations) | 1 | 0
Meningitis Viral (Infections and infestations) | 0 | 1
Nasal Abscess (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 3 | 1
Osteomyelitis (Infections and infestations) | 6 | 4
Otitis Externa (Infections and infestations) | 2 | 0
Otitis Media (Infections and infestations) | 1 | 1
Otitis Media Chronic (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic Abscess (Infections and infestations) | 1 | 0
Peridiverticular Abscess (Infections and infestations) | 0 | 1
Perihepatic Abscess (Infections and infestations) | 1 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0
Peritoneal Abscess (Infections and infestations) | 1 | 0
Peritonsillar Abscess (Infections and infestations) | 2 | 0
Periumbilical Abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 157 | 197
Pneumonia Bacterial (Infections and infestations) | 5 | 6
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Post Procedural Cellulitis (Infections and infestations) | 1 | 0
Post Procedural Infection (Infections and infestations) | 5 | 2
Postoperative Wound Infection (Infections and infestations) | 5 | 2
Pulmonary Tuberculosis (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 3 | 4
Pyelonephritis Acute (Infections and infestations) | 4 | 4
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Pyoderma (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1
Rectal Abscess (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 8 | 9
Salmonellosis (Infections and infestations) | 0 | 2
Scrotal Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 28 | 29
Septic Shock (Infections and infestations) | 11 | 7
Sialoadenitis (Infections and infestations) | 1 | 0
Skin Bacterial Infection (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 3
Streptococcal Bacteraemia (Infections and infestations) | 0 | 2
Streptococcal Sepsis (Infections and infestations) | 1 | 0
Subacute Endocarditis (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 3
Syphilis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 4
Tuberculosis (Infections and infestations) | 0 | 1
Tuberculous Pleurisy (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 12
Urinary Tract Infection (Infections and infestations) | 35 | 47
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1
Urinary Tract Infection Staphylococcal (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 8 | 11
Varicella (Infections and infestations) | 0 | 1
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 2 | 2
Viral Labyrinthitis (Infections and infestations) | 1 | 0
West Nile Viral Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 3 | 5
Wound Sepsis (Infections and infestations) | 1 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 2 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 5 | 6
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 | 0
Back Injury (Injury, poisoning and procedural complications) | 0 | 1
Brain Contusion (Injury, poisoning and procedural complications) | 0 | 1
Burns Third Degree (Injury, poisoning and procedural complications) | 1 | 1
Carbon Monoxide Poisoning (Injury, poisoning and procedural complications) | 1 | 1
Cardiac Valve Rupture (Injury, poisoning and procedural complications) | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 2
Chest Injury (Injury, poisoning and procedural complications) | 2 | 2
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 2
Compression Fracture (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 4 | 6
Drug Toxicity (Injury, poisoning and procedural complications) | 0 | 1
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 | 1
Face Injury (Injury, poisoning and procedural complications) | 0 | 2
Facial Bones Fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 15 | 11
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 10 | 15
Femur Fracture (Injury, poisoning and procedural complications) | 10 | 14
Fibula Fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 1
Head Injury (Injury, poisoning and procedural complications) | 8 | 6
Hip Fracture (Injury, poisoning and procedural complications) | 15 | 16
Humerus Fracture (Injury, poisoning and procedural complications) | 7 | 5
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 3
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 2 | 2
Injury (Injury, poisoning and procedural complications) | 1 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 5 | 2
Joint Injury (Injury, poisoning and procedural complications) | 0 | 3
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 | 2
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 3 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 3
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1
Neck Injury (Injury, poisoning and procedural complications) | 1 | 0
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1 | 9
Overdose (Injury, poisoning and procedural complications) | 4 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 2
Pelvic Fracture (Injury, poisoning and procedural complications) | 3 | 3
Periorbital Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 2 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 11 | 10
Postoperative Respiratory Distress (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 4
Radius Fracture (Injury, poisoning and procedural complications) | 3 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 6 | 12
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skeletal Injury (Injury, poisoning and procedural complications) | 2 | 0
Skin Injury (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 4
Skull Fractured Base (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Column Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 3 | 6
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 2
Splenic Rupture (Injury, poisoning and procedural complications) | 0 | 2
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 2 | 2
Subdural Haematoma (Injury, poisoning and procedural complications) | 15 | 16
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 2 | 6
Tendon Rupture (Injury, poisoning and procedural complications) | 2 | 0
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 8 | 4
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 2
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 4
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 3 | 3
Traumatic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 2 | 2
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 3 | 5
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wound Haemorrhage (Injury, poisoning and procedural complications) | 3 | 6
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 7 | 2
Arteriogram (Investigations) | 1 | 0
Arteriogram Coronary (Investigations) | 0 | 3
Aspartate Aminotransferase Increased (Investigations) | 5 | 1
Bilirubin Conjugated Increased (Investigations) | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Blood Amylase Increased (Investigations) | 0 | 1
Blood Bilirubin Increased (Investigations) | 4 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Blood Glucose Increased (Investigations) | 1 | 1
Blood Potassium Decreased (Investigations) | 0 | 1
Blood Pressure Increased (Investigations) | 2 | 4
C-Reactive Protein Increased (Investigations) | 0 | 1
Chest X-Ray Abnormal (Investigations) | 0 | 1
Coagulation Time Prolonged (Investigations) | 0 | 1
Dexamethasone Suppression Test Positive (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 1
Heart Rate Decreased (Investigations) | 1 | 1
Heart Rate Increased (Investigations) | 0 | 1
Heart Rate Irregular (Investigations) | 1 | 0
Hepatic Enzyme Abnormal (Investigations) | 0 | 2
Hepatic Enzyme Increased (Investigations) | 8 | 13
International Normalised Ratio Abnormal (Investigations) | 0 | 2
International Normalised Ratio Increased (Investigations) | 16 | 23
Intraocular Pressure Increased (Investigations) | 1 | 0
Laboratory Test Interference (Investigations) | 0 | 1
Lipase Increased (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 10 | 14
Occult Blood (Investigations) | 1 | 2
Occult Blood Positive (Investigations) | 1 | 1
Pancreatic Enzymes Increased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 1 | 2
Weight Decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 18 | 16
Diabetes Mellitus (Metabolism and nutrition disorders) | 32 | 23
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 9 | 8
Diabetic Foot (Metabolism and nutrition disorders) | 5 | 4
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 6 | 4
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperosmolar State (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 19 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 3
Neuroglycopenia (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Podagra (Metabolism and nutrition disorders) | 0 | 1
Shock Hypoglycaemic (Metabolism and nutrition disorders) | 0 | 2
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 6 | 5
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 13
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture Nonunion (Musculoskeletal and connective tissue disorders) | 2 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 9 | 10
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 5 | 4
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 2
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29 | 48
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 2
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Soft Tissue Haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 5
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2
Sympathetic Posterior Cervical Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8
Benign Colonic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Neoplasm of Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Neoplasm of Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Bladder Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Brain Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 15
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 14
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Colon Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0
Endometrial Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epiglottic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Gastric Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Infected Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intra-Abdominal Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large Cell Carcinoma of the Respiratory Tract Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo Maligna Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 10
Lung Squamous Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Malignant Palate Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Urinary Tract Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Mesothelioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Metastases to Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Carcinoma of the Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neurilemmoma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Non-Hodgkin's Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Paraneoplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 16
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 3
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Rectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Ureteric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anoxic Encephalopathy (Nervous system disorders) | 1 | 3
Aphasia (Nervous system disorders) | 2 | 1
Balance Disorder (Nervous system disorders) | 0 | 2
Basal Ganglia Haemorrhage (Nervous system disorders) | 2 | 0
Brachial Plexopathy (Nervous system disorders) | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1
Brain Stem Infarction (Nervous system disorders) | 0 | 1
Carotid Arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid Artery Disease (Nervous system disorders) | 1 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 1
Carotid Artery Stenosis (Nervous system disorders) | 5 | 6
Carpal Tunnel Syndrome (Nervous system disorders) | 2 | 1
Cauda Equina Syndrome (Nervous system disorders) | 1 | 0
Central Pain Syndrome (Nervous system disorders) | 0 | 1
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 2
Cerebral Arteriosclerosis (Nervous system disorders) | 3 | 0
Cerebral Haematoma (Nervous system disorders) | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 7 | 9
Cerebral Infarction (Nervous system disorders) | 2 | 2
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 14 | 8
Cerebrovascular Disorder (Nervous system disorders) | 1 | 1
Cerebrovascular Insufficiency (Nervous system disorders) | 1 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 1
Chorea (Nervous system disorders) | 0 | 1
Clonic Convulsion (Nervous system disorders) | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Complex Partial Seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 11 | 12
Dementia (Nervous system disorders) | 3 | 5
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 1
Diabetic Autonomic Neuropathy (Nervous system disorders) | 0 | 1
Diabetic Neuropathy (Nervous system disorders) | 3 | 9
Dizziness (Nervous system disorders) | 4 | 4
Dysarthria (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 3 | 3
Epilepsy (Nervous system disorders) | 11 | 12
Facial Palsy (Nervous system disorders) | 0 | 1
Facial Paresis (Nervous system disorders) | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 2 | 2
Haemorrhage Intracranial (Nervous system disorders) | 13 | 34
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 1 | 2
Haemorrhagic Stroke (Nervous system disorders) | 16 | 14
Haemorrhagic Transformation Stroke (Nervous system disorders) | 6 | 11
Headache (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 1 | 1
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0
Hypoxic Encephalopathy (Nervous system disorders) | 0 | 3
Iiird Nerve Paralysis (Nervous system disorders) | 0 | 1
Intercostal Neuralgia (Nervous system disorders) | 0 | 2
Intracranial Aneurysm (Nervous system disorders) | 0 | 1
Intracranial Haematoma (Nervous system disorders) | 1 | 2
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic Neuropathy (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 18 | 26
Lacunar Infarction (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 1 | 1
Lumbar Radiculopathy (Nervous system disorders) | 1 | 1
Metabolic Encephalopathy (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 0 | 1
Myasthenia Gravis (Nervous system disorders) | 1 | 0
Nerve Compression (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 3 | 1
Parkinson's Disease (Nervous system disorders) | 2 | 3
Parkinsonism (Nervous system disorders) | 1 | 1
Partial Seizures (Nervous system disorders) | 2 | 1
Partial Seizures with Secondary Generalisation (Nervous system disorders) | 1 | 0
Petit Mal Epilepsy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 2 | 1
Postictal Paralysis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 6 | 5
Radicular Syndrome (Nervous system disorders) | 1 | 0
Radiculitis (Nervous system disorders) | 0 | 1
Radiculitis Lumbosacral (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 4 | 4
Senile Dementia (Nervous system disorders) | 1 | 0
Sensory Disturbance (Nervous system disorders) | 1 | 0
Simple Partial Seizures (Nervous system disorders) | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 4 | 5
Syncope (Nervous system disorders) | 55 | 42
Toxic Encephalopathy (Nervous system disorders) | 0 | 1
Transient Global Amnesia (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 50 | 71
Vascular Dementia (Nervous system disorders) | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 5 | 3
Vertebrobasilar Insufficiency (Nervous system disorders) | 6 | 4
Vith Nerve Disorder (Nervous system disorders) | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute Psychosis (Psychiatric disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Alcohol Abuse (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Completed Suicide (Psychiatric disorders) | 1 | 2
Confusional State (Psychiatric disorders) | 4 | 5
Delirium (Psychiatric disorders) | 2 | 1
Delusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 9
Disorientation (Psychiatric disorders) | 1 | 1
Generalised Anxiety Disorder (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 2
Hallucination, Visual (Psychiatric disorders) | 1 | 0
Mental Disorder Due to A General Medical Condition (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 3 | 4
Mood Disorder Due to A General Medical Condition (Psychiatric disorders) | 1 | 0
Neurosis (Psychiatric disorders) | 0 | 1
Panic Disorder (Psychiatric disorders) | 0 | 2
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 1
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1
Bladder Prolapse (Renal and urinary disorders) | 1 | 0
Calculus Bladder (Renal and urinary disorders) | 4 | 1
Calculus Ureteric (Renal and urinary disorders) | 2 | 3
Calculus Urethral (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 1
Cystitis Erosive (Renal and urinary disorders) | 1 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0
Focal Segmental Glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 62 | 46
Haemorrhage Urinary Tract (Renal and urinary disorders) | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Hypertensive Nephropathy (Renal and urinary disorders) | 0 | 1
Kidney Enlargement (Renal and urinary disorders) | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 9 | 9
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 2 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 0 | 1
Obstructive Uropathy (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal Artery Arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 1
Renal Colic (Renal and urinary disorders) | 1 | 3
Renal Cyst (Renal and urinary disorders) | 1 | 2
Renal Failure (Renal and urinary disorders) | 27 | 18
Renal Failure Acute (Renal and urinary disorders) | 37 | 46
Renal Failure Chronic (Renal and urinary disorders) | 9 | 8
Renal Haemorrhage (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 5 | 8
Ureteric Haemorrhage (Renal and urinary disorders) | 0 | 2
Urethral Haemorrhage (Renal and urinary disorders) | 2 | 0
Urethral Stenosis (Renal and urinary disorders) | 5 | 2
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 0 | 2
Urinary Bladder Polyp (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 2 | 1
Urinary Retention (Renal and urinary disorders) | 12 | 7
Urinary Tract Obstruction (Renal and urinary disorders) | 2 | 0
Urogenital Haemorrhage (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 15 | 15
Endometrial Hyperplasia (Reproductive system and breast disorders) | 2 | 1
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 3 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 | 0
Genital Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 4 | 3
Oedema Genital (Reproductive system and breast disorders) | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 2 | 2
Prostatic Obstruction (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Scrotal Oedema (Reproductive system and breast disorders) | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 2 | 1
Uterine Polyp (Reproductive system and breast disorders) | 4 | 2
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 6 | 2
Vulval Ulceration (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Brain Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 59 | 56
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diaphragmatic Hernia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 25
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 | 41
Foreign Body Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Laryngeal Polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Mediastinal Haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal Cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary Amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 15 | 18
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Microemboli (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 | 18
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 2
Dry Gangrene (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 5
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 2 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 5 | 8
Skin Ulcer Haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 2
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Umbilical Haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria Chronic (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac Pacemaker Battery Replacement (Surgical and medical procedures) | 0 | 2
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 3 | 1
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 3 | 2
Cardiac Pacemaker Revision (Surgical and medical procedures) | 0 | 1
Cardioversion (Surgical and medical procedures) | 0 | 1
Carpal Tunnel Decompression (Surgical and medical procedures) | 1 | 1
Cataract Operation (Surgical and medical procedures) | 2 | 1
Finger Amputation (Surgical and medical procedures) | 2 | 0
Foot Amputation (Surgical and medical procedures) | 1 | 0
Haemorrhoid Operation (Surgical and medical procedures) | 1 | 0
Hip Arthroplasty (Surgical and medical procedures) | 3 | 1
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 | 1
Inguinal Hernia Repair (Surgical and medical procedures) | 2 | 0
Knee Arthroplasty (Surgical and medical procedures) | 1 | 1
Knee Operation (Surgical and medical procedures) | 0 | 1
Limb Operation (Surgical and medical procedures) | 1 | 0
Penile Repair (Surgical and medical procedures) | 1 | 0
Percutaneous Coronary Intervention (Surgical and medical procedures) | 2 | 0
Polypectomy (Surgical and medical procedures) | 1 | 1
Prostatectomy (Surgical and medical procedures) | 0 | 1
Skin Graft (Surgical and medical procedures) | 0 | 1
Skin Neoplasm Excision (Surgical and medical procedures) | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 3 | 1
Transurethral Prostatectomy (Surgical and medical procedures) | 2 | 0
Varicose Vein Operation (Surgical and medical procedures) | 0 | 1
Wound Drainage (Surgical and medical procedures) | 1 | 0
Accelerated Hypertension (Vascular disorders) | 1 | 0
Angiopathy (Vascular disorders) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 6 | 7
Aortic Aneurysm Rupture (Vascular disorders) | 2 | 6
Aortic Dilatation (Vascular disorders) | 1 | 0
Aortic Disorder (Vascular disorders) | 0 | 1
Aortic Dissection (Vascular disorders) | 1 | 2
Aortic Stenosis (Vascular disorders) | 1 | 0
Arterial Occlusive Disease (Vascular disorders) | 1 | 2
Arterial Stenosis Limb (Vascular disorders) | 2 | 0
Arterial Thrombosis Limb (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 2 | 2
Arteriosclerosis Obliterans (Vascular disorders) | 4 | 3
Arteriovenous Fistula (Vascular disorders) | 0 | 1
Bleeding Varicose Vein (Vascular disorders) | 4 | 1
Circulatory Collapse (Vascular disorders) | 3 | 1
Deep Vein Thrombosis (Vascular disorders) | 12 | 15
Diabetic Vascular Disorder (Vascular disorders) | 1 | 1
Diastolic Hypertension (Vascular disorders) | 0 | 1
Essential Hypertension (Vascular disorders) | 0 | 2
Extremity Necrosis (Vascular disorders) | 2 | 1
Femoral Arterial Stenosis (Vascular disorders) | 1 | 1
Femoral Artery Occlusion (Vascular disorders) | 1 | 2
Haematoma (Vascular disorders) | 32 | 42
Haemodynamic Instability (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 5
Haemorrhagic Infarction (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 26 | 28
Hypertensive Crisis (Vascular disorders) | 16 | 16
Hypertensive Emergency (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 13 | 15
Hypovolaemic Shock (Vascular disorders) | 4 | 2
Intermittent Claudication (Vascular disorders) | 2 | 0
Jugular Vein Distension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Microangiopathy (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 4 | 8
Peripheral Arterial Occlusive Disease (Vascular disorders) | 8 | 8
Peripheral Ischaemia (Vascular disorders) | 10 | 2
Peripheral Vascular Disorder (Vascular disorders) | 7 | 3
Phlebitis (Vascular disorders) | 1 | 1
Raynaud's Phenomenon (Vascular disorders) | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis Migrans (Vascular disorders) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 3
Varicose Ulceration (Vascular disorders) | 0 | 1
Varicose Vein (Vascular disorders) | 3 | 2
Vasculitis (Vascular disorders) | 0 | 1
Vasculitis Necrotising (Vascular disorders) | 1 | 0
Venous Insufficiency (Vascular disorders) | 0 | 2
Venous Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 2
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Splenic Haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Chronotropic Incompetence (Cardiac disorders) | 1 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0
Mitral Valve Stenosis (Cardiac disorders) | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1
External Ear Disorder (Ear and labyrinth disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Barrett's Oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 1 | 0
Peritoneal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Feeling Abnormal (General disorders) | 0 | 1
Implant Site Effusion (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0
Acute Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Haemorrhagic Hepatic Cyst (Hepatobiliary disorders) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 1
Haemophilus Infection (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Pharyngeal Abscess (Infections and infestations) | 0 | 1
Pseudomembranous Colitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 1
Sepsis Syndrome (Infections and infestations) | 0 | 1
Cardiac Function Disturbance Postoperative (Injury, poisoning and procedural complications) | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1
Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 1
Venous Injury (Injury, poisoning and procedural complications) | 1 | 0
Aspiration Bronchial (Investigations) | 0 | 1
Prothrombin Level Decreased (Investigations) | 0 | 1
Prothrombin Time Prolonged (Investigations) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Soft Tissue Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mediastinum Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory Anaemia with An Excess of Blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteral Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar Atrophy (Nervous system disorders) | 1 | 0
Diabetic Hyperosmolar Coma (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 1 | 0
Prostatic Atrophy (Reproductive system and breast disorders) | 0 | 1
Prostatic Intraepithelial Neoplasia (Reproductive system and breast disorders) | 0 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal Hernia Repair (Surgical and medical procedures) | 0 | 1
Colostomy Closure (Surgical and medical procedures) | 1 | 0
Ileostomy (Surgical and medical procedures) | 1 | 0
Malignant Tumour Excision (Surgical and medical procedures) | 1 | 0
Lymphatic Fistula (Vascular disorders) | 1 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 0 | 1
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=7111) | Warfarin (N=7125)
Diarrhoea (Gastrointestinal disorders) | 384 | 401
Oedema Peripheral (General disorders) | 443 | 451
Bronchitis (Infections and infestations) | 377 | 401
Nasopharyngitis (Infections and infestations) | 430 | 464
Dizziness (Nervous system disorders) | 445 | 453
Headache (Nervous system disorders) | 332 | 367
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 389 | 382
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 705 | 594
Cough (Respiratory, thoracic and mediastinal disorders) | 356 | 363

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less